CLINICAL TRIAL: NCT03481556
Title: An Open-Label Phase 1/2a Study of the Safety and Efficacy of Melflufen and Dexamethasone in Combination With Either Bortezomib or Daratumumab in Patients With Relapsed or Relapsed-Refractory Multiple Myeloma
Brief Title: Study of Melphalan Flufenamide (Melflufen) + Dex With Bortezomib or Daratumumab in Patients With RRMM
Acronym: ANCHOR
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study following an FDA request of a partial clinical hold.
Sponsor: Oncopeptides AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP-104
Record Dates: First submitted 2018-03-06; First posted 2018-03-29 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — L-melphalanyl-p-L-fluorophenylalanine ethyl ester; melflufen; Dexamethasone; dexamethasone acetate; Calcium Dobesilate; Bortezomib; daratumumab; darlin protein, Dictyostelium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A (melflufen+bortezomib+dex) (Experimental): Melflufen 30 mg and 40 mg or 20 mg i.v. Day 1 of each 28-day cycle in combination with bortezomib at 1.3mg/m² S.Q. on Days 1, 4, 8, 11 and dexamethasone 20 mg (12 mg ≥ 75 years) Days 1, 4, 8, 11 and 40 mg (20 mg ≥ 75 years) on Day 15 and 22 of each 28-day cycle.
  Interventions: Drug: Melphalan flufenamide (Melflufen); Drug: Dexamethasone; Drug: Bortezomib
- B (melflufen+daratumumab+dex) (Experimental): Melflufen 30 mg and 40 mg or 20 mg i.v. Day 1 of each 28-day cycle in combination with daratumumab 16 mg/kg weekly for 8 doses, every other week for 8 doses and then once every 4 weeks. Dexamethasone p.o. 40 mg weekly (20 mg weekly for patients age ≥ 75 years).
  Interventions: Drug: Melphalan flufenamide (Melflufen); Drug: Dexamethasone; Drug: Daratumumab

INTERVENTIONS:
Drug: Melphalan flufenamide (Melflufen) — Intravenous infusion
Drug: Dexamethasone — Oral tablets
  Other Names: Dex; Fortecortin; Decadron
Drug: Bortezomib — Subcutaneous administration
  Other Names: Velcade
  Arms: A (melflufen+bortezomib+dex)
Drug: Daratumumab — Intravenous infusion
  Other Names: Dara; Darzalex
  Arms: B (melflufen+daratumumab+dex)

SUMMARY:
This is an open-label Phase 1/2a study which will enroll patients that have relapsed or relapsed-refractory multiple myeloma to combination regimens of melflufen with currently approved agents. Patients will receive either melflufen+dexamethasone+bortezomib or melflufen+dexamethasone+daratumumab.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older
2. A prior diagnosis of multiple myeloma with documented disease progression in need of treatment at time of screening
3. One to four prior lines of therapy
4. Measurable disease defined as any of the following:

   * Serum monoclonal protein ≥ 0.5 g/dL by serum protein electrophoresis (SPEP)
   * ≥ 200 mg/24 hours of monoclonal protein in the urine on 24-hour urine electrophoresis (UPEP)
   * Serum free light chain (SFLC) ≥ 10 mg/dL AND abnormal serum kappa to lambda free light chain ratio
5. Life expectancy of ≥ 6 months
6. ECOG performance status ≤ 2. (Patients with lower performance status based solely on bone pain secondary to multiple myeloma may be eligible following consultation and approval of the medical monitor)
7. Patient is a female of childbearing potential (FCBP)* with a negative serum or urine pregnancy test prior to initiation of therapy and agrees to practice appropriate methods of birth control, or the patient is male and agrees to practice appropriate methods of birth control
8. Ability to understand the purpose and risks of the study and provide signed and dated informed consent
9. 12-lead Electrocardiogram (ECG) with QT interval calculated by Fridericia Formula (QTcF) interval of ≤ 470 msec
10. Adequate organ function with the following laboratory results during screening (within 21 days) and immediately before study drug administration on Cycle 1 Day 1:

    * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3 (1.0 x 109/L) (Growth factors cannot be used within 10 days (14 days for pegfilgrastim) prior to initiation of therapy)
    * Platelet count ≥ 75,000 cells/mm3 (75 x 109/L) (without required transfusions during the 10 days prior to initiation of therapy)
    * Hemoglobin ≥ 8.0 g/dl (red blood cell (RBC) transfusions are permitted)
    * Total Bilirubin ≤ 1.5 x upper limit of normal (ULN), or patients diagnosed with Gilbert's syndrome, that have been reviewed and approved by the medical monitor
    * AST/SGOT and ALT/SGPT ≤ 3.0 x ULN
    * Renal function: Estimated creatinine clearance by Cockcroft-Gault formula ≥ 45 mL/min and serum creatinine ≤ 2 mg/dL
11. Must have, or be willing to have an acceptable central catheter. (Port a cath, peripherally inserted central catheter [PICC] line, or central venous catheter)

    Regimen A
12. Must be intolerant or refractory to a prior IMiD; refractory defined as failure to respond (MR or better) or progression while on therapy or within 60 days of last dose.

    Regimen B
13. Must have had a prior IMiD and a proteasome inhibitor (PI); alone or in combination and must be refractory or intolerant to an IMiD, PI or both.

    * (FCBP) is any sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (not having menstrual cycles due to cancer therapy does not rule out childbearing potential) for at least 24 consecutive months.

Exclusion Criteria:

1. Primary refractory disease (i.e. never responded with ≥ MR to any prior therapy)
2. Evidence of mucosal or internal bleeding and/or are platelet transfusion refractory (i.e. platelet count fails to increase by > 10,000 cells/mm3 after transfusion of an appropriate dose of platelets)
3. Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient or would adversely affect his/her participating in this study. Examples of such conditions are: a significant history of cardiovascular disease (e.g., myocardial infarction, significant conduction system abnormalities, uncontrolled hypertension, ≥ Grade 3 thromboembolic event in the last 6 months)
4. Known active infection requiring parenteral or oral anti-infective treatment within 14 days of initiation of therapy
5. Other malignancy diagnosed or requiring treatment within the past 3 years with the exception of adequately treated basal cell carcinoma, squamous cell skin cancer, carcinoma in-situ of the cervix or breast or very low and low risk prostate cancer in active surveillance
6. Pregnant or breast-feeding females
7. Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse compliance or follow-up evaluation
8. Known human immunodeficiency virus or active hepatitis B or C viral infection
9. Concurrent symptomatic amyloidosis or plasma cell leukemia
10. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes)
11. Previous cytotoxic therapies, including cytotoxic investigational agents, for multiple myeloma within 3 weeks (6 weeks for nitrosoureas) prior to initiation of therapy. The use of live vaccines within 30 days before initiation of therapy. IMiDs, PIs and or corticosteroids within 2 weeks prior to initiation of therapy. Other investigational therapies and monoclonal antibodies (mAb) within 4 weeks of initiation of therapy Prednisone up to but no more than 10 mg orally once daily (q.d.) or its equivalent for symptom management of comorbid conditions is permitted but dose should be stable for at least 7 days prior to initiation of therapy
12. Residual side effects to previous therapy > Grade 1 prior to initiation of therapy (Alopecia any grade and/or neuropathy Grade 1 without pain are permitted)
13. Prior peripheral stem cell transplant within 12 weeks of initiation of therapy
14. Prior allogeneic stem cell transplantation with active graft-versus-host- disease
15. Prior major surgical procedure or radiation therapy within 4 weeks of initiation of therapy (this does not include limited course of radiation used for management of bone pain within 7 days of initiation of therapy)
16. Known intolerance to the required dose and schedule of steroid therapy as determined by the investigator
17. Prior treatment with melflufen

    Regimen A
18. Refractory to a PI in the last line of therapy prior to enrollment in this trial; refractory defined as failure to respond (MR or better) or progression while on therapy or within 60 days of last dose
19. History of allergic reaction/hypersensitivity attributed to compounds containing boron, mannitol, polysorbate 80 or sodium citrate dihydrate

    Regimen B
20. Prior exposure to an antiCD-38 mAb
21. Chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) less than 50% of predicted normal
22. Moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification
23. ≥ Grade 3 conduction system abnormalities unless patient has a pacemaker
24. Active hepatitis B (defined as HBsAg+) or those at risk for reactivation (HBsAg-, Anti- HBs+, Anti-HBc+)

    * Patients with prior hepatitis B vaccine are permitted (defined as HBsAg-, Anti-HBs+, Anti-HBc-)

      * Non-active hepatitis B (HBsAg-, Anti-HBs+, Anti-HBc+) may only be enrolled after approval of the sponsor and consideration of risk of reactivation (additional screening and monitoring for reactivation of Hepatitis B and consultation with a liver disease specialist may be required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - The Ohio State University, Columbus, Ohio
- Czechia (4):
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice Hradec Králové, Hradec Králové
  - Fakultní nemocnice Ostrava, Ostrava
  - Všeobecná fakultní nemocnice, Prague
- France (5):
  - Hôpital Morvan, Brest
  - Centre Jean Bernard - Clinique Victor Hugo, Le Mans
  - Hôpital privé du Confluent, Nantes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire Institut Gustave Roussy, Villejuif
- Spain (5):
  - Hospital Universitai Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Hospitalario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 56 participants were enrolled across 13 sites in the Czech Republic, France, Spain and the United States.
Pre-assignment Details: A total of 56 participants were enrolled in the study, all of whom received study treatment.
Groups:
- Regimen A - Melflufen 30mg + Bortezomib + Dexamethasone: Participants were administered intravenous (IV) melflufen at a dose of 30 mg on Day 1 of each 28-day cycle in combination with subcutaneous (SQ) bortezomib at a dose of 1.3mg/m^2 on Days 1, 4, 8, and 11 and dexamethasone orally (PO) at a dose of 20 mg (12 mg if the participants is ≥ 75 years of age) on Days 1, 4, 8, and 11 and 40 mg (20 mg if the participants is ≥ 75 years of age) on Day 15 and 22 of each 28-day cycle.
- Regimen A - Melflufen 40mg + Bortezomib + Dexamethasone: Participants were administered intravenous (IV) melflufen at a dose of 40 mg on Day 1 of each 28-day cycle in combination with subcutaneous (SQ) bortezomib at a dose of 1.3mg/m^2 on Days 1, 4, 8, and 11 and dexamethasone orally (PO) at a dose of 20 mg (12 mg if the participants is ≥ 75 years of age) on Days 1, 4, 8, and 11 and 40 mg (20 mg if the participants is ≥ 75 years of age) on Day 15 and 22 of each 28-day cycle.
- Regimen B - Melflufen 30mg + Daratumumab + Dexamethasone: Participants were administered intravenous (IV) melflufen at a dose of 30 mg on Day 1 of each 28-day cycle in combination with IV daratumumab at a dose of 16 mg/kg weekly for 8 doses, every other week for 8 doses and then once every 4 weeks. Participants were also administered dexamethasone orally (PO) at a dose of 40 mg weekly (20 mg weekly if the participants is ≥ 75 years of age).
- Regimen B - Melflufen 40mg + Daratumumab + Dexamethasone: Participants were administered intravenous (IV) melflufen at a dose of 40 mg on Day 1 of each 28-day cycle in combination with IV daratumumab at a dose of 16 mg/kg weekly for 8 doses, every other week for 8 doses and then once every 4 weeks. Participants were also administered dexamethasone orally (PO) at a dose of 40 mg weekly (20 mg weekly if the participants is ≥ 75 years of age).
Period: Overall Study
Arm/Group | Regimen A - Melflufen 30mg + Bortezomib + Dexamethasone | Regimen A - Melflufen 40mg + Bortezomib + Dexamethasone | Regimen B - Melflufen 30mg + Daratumumab + Dexamethasone | Regimen B - Melflufen 40mg + Daratumumab + Dexamethasone
Started | 15 | 8 | 6 | 27
Completed | 0 | 1 | 1 | 2
Not Completed | 15 | 7 | 5 | 25
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 4 | 2 | 3 | 16
Not completed — Study Terminated by Sponsor | 10 | 5 | 2 | 9

BASELINE CHARACTERISTICS:
Population: Participants included in the Safety Analysis Set were included in the Baseline Characteristics. The Safety Analysis Set includes all patients that have received at least 1 dose (or partial dose) of melflufen, dexamethasone, or partner therapy (bortezomib or daratumumab).
Groups:
- Regimen A - Melflufen 30mg + Bortezomib + Dexamethasone: Participants were administered IV melflufen at a dose of 30 mg on Day 1 of each 28-day cycle in combination with SQ bortezomib at a dose of 1.3mg/m^2 on Days 1, 4, 8, and 11 and dexamethasone PO at a dose of 20 mg (12 mg if the participants is ≥ 75 years of age) on Days 1, 4, 8, and 11 and 40 mg (20 mg if the participants is ≥ 75 years of age) on Day 15 and 22 of each 28-day cycle.
- Regimen A - Melflufen 40mg + Bortezomib + Dexamethasone: Participants were administered IV melflufen at a dose of 40 mg on Day 1 of each 28-day cycle in combination with SQ bortezomib at a dose of 1.3mg/m^2 on Days 1, 4, 8, and 11 and dexamethasone PO at a dose of 20 mg (12 mg if the participants is ≥ 75 years of age) on Days 1, 4, 8, and 11 and 40 mg (20 mg if the participants is ≥ 75 years of age) on Day 15 and 22 of each 28-day cycle.
- Regimen B - Melflufen 30mg + Daratumumab + Dexamethasone: Participants were administered IV melflufen at a dose of 30 mg on Day 1 of each 28-day cycle in combination with IV daratumumab at a dose of 16 mg/kg weekly for 8 doses, every other week for 8 doses and then once every 4 weeks. Participants were also administered dexamethasone orally (PO) at a dose of 40 mg weekly (20 mg weekly if the participants is ≥ 75 years of age).
- Regimen B - Melflufen 40mg + Daratumumab + Dexamethasone: Participants were administered IV melflufen at a dose of 40 mg on Day 1 of each 28-day cycle in combination with IV daratumumab at a dose of 16 mg/kg weekly for 8 doses, every other week for 8 doses and then once every 4 weeks. Participants were also administered dexamethasone orally (PO) at a dose of 40 mg weekly (20 mg weekly if the participants is ≥ 75 years of age).
- Total: Total of all reporting groups
Arm/Group | Regimen A - Melflufen 30mg + Bortezomib + Dexamethasone | Regimen A - Melflufen 40mg + Bortezomib + Dexamethasone | Regimen B - Melflufen 30mg + Daratumumab + Dexamethasone | Regimen B - Melflufen 40mg + Daratumumab + Dexamethasone | Total
Number analyzed (Participants) | 15 | 8 | 6 | 27 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (8.17) | 69.4 (5.13) | 60.5 (12.13) | 62.3 (11.15) | 65.1 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 3 | 8 | 19
  Male | 8 | 7 | 3 | 19 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 14 | 8 | 6 | 23 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 15 | 8 | 6 | 21 | 50
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Description: Toxicity was graded according to the National Cancer Institute - Common Terminology Criteria for Adverse Events Version 4.03.
  DLT criteria that apply to Regimens A and B:
  * Grade 3 non-hematologic toxicity preventing the administration of > 1 dose of bortezomib or daratumumab during the 1st cycle.
  * Grade 4 or greater non-hematologic toxicity.
  * Grade 4 thrombocytopenia (platelet count < 25,000 cells/ mm^3) preventing the administration of > 1 dose of bortezomib or daratumumab during the 1st cycle or with clinically significant bleeding during the 1st cycle.
  * Grade 4 neutropenia (ANC < 500 cells/mm^3), lasting more than 7 days during the 1st cycle.
  * Greater than 14 days' delay to meet the criteria for the start of a new cycle (Cycle 2) due to toxicity.
Time Frame: Cycle 1: Day 1 to Day 28
Population: Only participants included in the DLT Analysis set were included in this analysis. The DLT Analysis Set was defined as all participants in Phase 1 that complete Cycle 1 of therapy or are discontinued due to a DLT event.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A - Melflufen 30mg + Bortezomib + Dexamethasone | Regimen A - Melflufen 40mg + Bortezomib + Dexamethasone | Regimen B - Melflufen 30mg + Daratumumab + Dexamethasone | Regimen B - Melflufen 40mg + Daratumumab + Dexamethasone
Number analyzed (Participants) | 6 | 6 | 3 | 6
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a best confirmed response of Partial Response (PR) or better.
Time Frame: Until disease progression, death or initiation of subsequent therapy (a maximum of 194.3 weeks)
Population: All participants included in the Safety Analysis Set were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Regimen A - Melflufen 30mg + Bortezomib + Dexamethasone | Regimen A - Melflufen 40mg + Bortezomib + Dexamethasone | Regimen B - Melflufen 30mg + Daratumumab + Dexamethasone | Regimen B - Melflufen 40mg + Daratumumab + Dexamethasone
Number analyzed (Participants) | 15 | 8 | 6 | 27
percentage of participants | 80 [51.9 to 95.7] | 75 [34.9 to 96.8] | 83.3 [35.9 to 99.6] | 70.4 [49.8 to 86.2]

3. Secondary Outcome: Best Response (BR)
Description: BR defined by International Myeloma Working Group Uniform Response Criteria. BR= Complete Response (CR)/Stringent CR (sCR) defined as below negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow/plus normal free light chain (FLC) ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence, Very Good Partial Response (VGPR)= serum and urine M-protein detectable by immunofixation but not on electrophoresis or > 90% reduction in serum M-protein plus urine M-protein level < 100 mg/24 hours, Partial Response (PR)= a > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by > 90% or to < 200 mg/24 hours, Minimal Response (MR), Stable Disease (SD)= not meeting the criteria for other response options, Progressive Disease (PD)= increase of > 25% from lowest response value in serum/urine M-component or bone marrow plasma cell percentage, or non-evaluable.
Time Frame: Until disease progression, death or initiation of subsequent therapy (a maximum of 194.3 weeks)
Population: All participants included in the Safety Analysis Set were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A - Melflufen 30mg + Bortezomib + Dexamethasone | Regimen A - Melflufen 40mg + Bortezomib + Dexamethasone | Regimen B - Melflufen 30mg + Daratumumab + Dexamethasone | Regimen B - Melflufen 40mg + Daratumumab + Dexamethasone
Number analyzed (Participants) | 15 | 8 | 6 | 27
Participants
  CR | 1 | 0 | 1 | 1
  sCR | 0 | 1 | 0 | 1
  VGPR | 2 | 3 | 2 | 6
  PR | 9 | 2 | 2 | 11
  MR | 1 | 0 | 0 | 1
  SD | 1 | 1 | 0 | 2
  PD | 0 | 0 | 0 | 1
  Non-evaluable | 0 | 0 | 0 | 0
  Missing | 1 | 1 | 1 | 4

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined for participants with confirmed objective response (PR or better, which includes PR, VGPR, CR and sCR) as the time from the first documentation of objective response to the first documentation of objective progression or to death due to any cause, whichever occurs first.
Time Frame: Until disease progression, death or initiation of subsequent therapy (a maximum of 194.3 weeks)
Population: Only participants included in the Safety Analysis Set who achieved a response of PR or better were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- A (Melflufen+Bortezomib+Dex) 30 mg: Participants were administered IV melflufen at a dose of 30 mg on Day 1 of each 28-day cycle in combination with SQ bortezomib at a dose of 1.3mg/m^2 on Days 1, 4, 8, and 11 and dexamethasone PO at a dose of 20 mg (12 mg if the participants is ≥ 75 years of age) on Days 1, 4, 8, and 11 and 40 mg (20 mg if the participants is ≥ 75 years of age) on Day 15 and 22 of each 28-day cycle.
- A (Melflufen+Bortezomib+Dex) 40 mg: Participants were administered IV melflufen at a dose of 40 mg on Day 1 of each 28-day cycle in combination with SQ bortezomib at a dose of 1.3mg/m^2 on Days 1, 4, 8, and 11 and dexamethasone PO at a dose of 20 mg (12 mg if the participants is ≥ 75 years of age) on Days 1, 4, 8, and 11 and 40 mg (20 mg if the participants is ≥ 75 years of age) on Day 15 and 22 of each 28-day cycle.
- B (Melflufen+Daratumumab+Dex) 30 mg: Participants were administered IV melflufen at a dose of 30 mg on Day 1 of each 28-day cycle in combination with IV daratumumab at a dose of 16 mg/kg weekly for 8 doses, every other week for 8 doses and then once every 4 weeks. Participants were also administered dexamethasone orally (PO) at a dose of 40 mg weekly (20 mg weekly if the participants is ≥ 75 years of age).
- B (Melflufen+Daratumumab+Dex) 40 mg: Participants were administered IV melflufen at a dose of 40 mg on Day 1 of each 28-day cycle in combination with IV daratumumab at a dose of 16 mg/kg weekly for 8 doses, every other week for 8 doses and then once every 4 weeks. Participants were also administered dexamethasone orally (PO) at a dose of 40 mg weekly (20 mg weekly if the participants is ≥ 75 years of age).
Arm/Group | A (Melflufen+Bortezomib+Dex) 30 mg | A (Melflufen+Bortezomib+Dex) 40 mg | B (Melflufen+Daratumumab+Dex) 30 mg | B (Melflufen+Daratumumab+Dex) 40 mg
Number analyzed (Participants) | 12 | 6 | 5 | 19
months | 9.0 [4.9 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | NA [NA to NA] — Median and confidence interval values could not be calculated as the fraction of participants experiencing events was too low. | 24.2 [10.60 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 9.9 [7.2 to 14.8]

5. Secondary Outcome: Time to Response (TTR)
Description: Time from Cycle 1 Day 1 to a response of PR or better.
Time Frame: Until disease progression, death or initiation of subsequent therapy (a maximum of 194.3 weeks)
Population: as for outcome 4
Measure: Median (Full Range); unit: months
Arm/Group | A (Melflufen+Bortezomib+Dex) 30 mg | A (Melflufen+Bortezomib+Dex) 40 mg | B (Melflufen+Daratumumab+Dex) 30 mg | B (Melflufen+Daratumumab+Dex) 40 mg
Number analyzed (Participants) | 12 | 6 | 5 | 19
months | 3.0 [1.0 to 8.6] | 2.2 [1.0 to 4.6] | 3.3 [1.0 to 4.2] | 1.1 [0.9 to 5.3]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time in months from date of initiation of therapy to the earlier of confirmed disease progression or death due to any cause.
Time Frame: Until disease progression, death or initiation of subsequent therapy (a maximum of 194.3 weeks)
Population: All participants included in the Safety Analysis Set were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A (Melflufen+Bortezomib+Dex) 30 mg | A (Melflufen+Bortezomib+Dex) 40 mg | B (Melflufen+Daratumumab+Dex) 30 mg | B (Melflufen+Daratumumab+Dex) 40 mg
Number analyzed (Participants) | 15 | 8 | 6 | 27
months | 10.0 [7.5 to 33.5] | 24.30 [2.90 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 28.4 [14.3 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 9.7 [6.7 to 14.2]

7. Secondary Outcome: Overall Survival (OS)
Description: Time from the first dose of melflufen to death due to any cause.
Time Frame: Up to 24 months following confirmed disease progression, or initiation of subsequent therapy (a maximum of 198.9 weeks)
Population: Only participants included in the Safety Analysis Set were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A (Melflufen+Bortezomib+Dex) 30 mg | A (Melflufen+Bortezomib+Dex) 40 mg | B (Melflufen+Daratumumab+Dex) 30 mg | B (Melflufen+Daratumumab+Dex) 40 mg
Number analyzed (Participants) | 15 | 8 | 6 | 27
months | 33.5 [9.00 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | NA [NA to NA] — Median and confidence interval values could not be calculated as the fraction of participants experiencing events was too low. | 35.0 [6.4 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 18.3 [14.29 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low.

8. Secondary Outcome: Duration of Clinical Benefit (DOCB)
Description: DOCB was defined as time in months from the first evidence of confirmed assessment of sCR, CR, VGPR, PR or MR to first confirmed disease progression, or to death due to any cause.
Time Frame: Until disease progression, death or initiation of subsequent therapy (a maximum of 194.3 weeks)
Population: All participants included in the Safety Analysis Set with a confirmed MR or better were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- B (Melflufen+Daratumumab+Dex) 30 mg: Participants were administered IV melflufen at a dose of 30 mg on Day 1 of each 28-day cycle in combination with daratumumab at a dose of 16 mg/kg weekly for 8 doses, every other week for 8 doses and then once every 4 weeks. Participants were also administered dexamethasone PO at a dose of 40 mg weekly (20 mg weekly if the participants is ≥ 75 years of age).
- B (Melflufen+Daratumumab+Dex) 40 mg: Participants were administered IV melflufen at a dose of 40 mg on Day 1 of each 28-day cycle in combination with daratumumab at a dose of 16 mg/kg weekly for 8 doses, every other week for 8 doses and then once every 4 weeks. Participants were also administered dexamethasone PO at a dose of 40 mg weekly (20 mg weekly if the participants is ≥ 75 years of age).
Arm/Group | A (Melflufen+Bortezomib+Dex) 30 mg | A (Melflufen+Bortezomib+Dex) 40 mg | B (Melflufen+Daratumumab+Dex) 30 mg | B (Melflufen+Daratumumab+Dex) 40 mg
Number analyzed (Participants) | 13 | 6 | 5 | 20
months | 15.7 [7.6 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 21.3 [13.7 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 27.20 [13.10 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 10.9 [8.40 to 14.50]

9. Secondary Outcome: Time to Progression (TTP)
Description: TTP defined as time from first dose to first documented confirmed progression.
Time Frame: Until disease progression, death or initiation of subsequent therapy (a maximum of 194.3 weeks)
Population: All participants in the Safety Analysis Set are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A (Melflufen+Bortezomib+Dex) 30 mg | A (Melflufen+Bortezomib+Dex) 40 mg | B (Melflufen+Daratumumab+Dex) 30 mg | B (Melflufen+Daratumumab+Dex) 40 mg
Number analyzed (Participants) | 15 | 8 | 6 | 27
months | 17.6 [7.5 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 24.3 [2.90 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 29.2 [14.3 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 11.5 [7.7 to 15.4]

10. Secondary Outcome: Clinical Benefit Rate (≥ Minimal Response)
Description: ≥ Minimal response for participants included sCR, CR, VGPR, PR and MR.
Time Frame: Until disease progression, death or initiation of subsequent therapy (a maximum of 194.3 weeks)
Population: All participants included in the Safety Analysis Set were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A (Melflufen+Bortezomib+Dex) 30 mg | A (Melflufen+Bortezomib+Dex) 40 mg | B (Melflufen+Daratumumab+Dex) 30 mg | B (Melflufen+Daratumumab+Dex) 40 mg
Number analyzed (Participants) | 15 | 8 | 6 | 27
percentage of participants | 86.7 [59.5 to 98.3] | 75.0 [34.9 to 96.8] | 83.3 [35.9 to 99.6] | 74.1 [53.7 to 88.9]

11. Secondary Outcome: Time to Next Treatment (TTNT)
Description: Defined as time from date of initiation of therapy to start of next line of therapy.
Time Frame: Until death or initiation of subsequent therapy (a maximum of 194.3 weeks)
Population: All participants included in the Safety Analysis Set were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A (Melflufen+Bortezomib+Dex) 30 mg | A (Melflufen+Bortezomib+Dex) 40 mg | B (Melflufen+Daratumumab+Dex) 30 mg | B (Melflufen+Daratumumab+Dex) 40 mg
Number analyzed (Participants) | 15 | 8 | 6 | 27
months | 33.50 [9.0 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 14.70 [3.90 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 26.25 [2.3 to NA] — Upper confidence interval value could not be calculated as the fraction of participants experiencing events was too low. | 9.5 [5.6 to 13.4]

12. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: TEAEs were defined as adverse events (AEs) that started after the first dose of study medication was administered and within 30 days of the last administration of the study treatment or before start of subsequent anticancer treatment (whichever occurred first) or that worsened after the first dose of study medication was administered.
Time Frame: Cycle 1 Day 1 up to a maximum of 198.9 weeks
Population: Only participants included in the Safety Analysis Set were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | A (Melflufen+Bortezomib+Dex) 30 mg | A (Melflufen+Bortezomib+Dex) 40 mg | B (Melflufen+Daratumumab+Dex) 30 mg | B (Melflufen+Daratumumab+Dex) 40 mg
Number analyzed (Participants) | 15 | 8 | 6 | 27
Participants
  Any TEAEs | 15 | 8 | 6 | 27
  Any Grade 3 or Higher TEAEs | 15 | 8 | 6 | 26

ADVERSE EVENTS:
Time Frame: Cycle 1 Day 1 up to a maximum of 198.9 weeks
Description: All AEs that were spontaneously reported by the participant or detected during or between visits by non-directive questioning, through physical examination, laboratory test, or other assessments were reported in the eCRF. All participants included in the Safety Analysis Set were included in this analysis.
Arm/Group | A (Melflufen+Bortezomib+Dex) 30 mg | A (Melflufen+Bortezomib+Dex) 40 mg | B (Melflufen+Daratumumab+Dex) 30 mg | B (Melflufen+Daratumumab+Dex) 40 mg
All-Cause Mortality (participants affected / at risk) | 4/15 | 2/8 | 3/6 | 16/27
Serious Adverse Events (participants affected / at risk) | 9/15 | 5/8 | 4/6 | 11/27
Other Adverse Events (participants affected / at risk) | 15/15 | 8/8 | 6/6 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A (Melflufen+Bortezomib+Dex) 30 mg (N=15) | A (Melflufen+Bortezomib+Dex) 40 mg (N=8) | B (Melflufen+Daratumumab+Dex) 30 mg (N=6) | B (Melflufen+Daratumumab+Dex) 40 mg (N=27)
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 3
COVID-19 pneumonia (Infections and infestations) | 2 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2
Infection (Infections and infestations) | 0 | 1 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0 | 1
Right ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A (Melflufen+Bortezomib+Dex) 30 mg (N=15) | A (Melflufen+Bortezomib+Dex) 40 mg (N=8) | B (Melflufen+Daratumumab+Dex) 30 mg (N=6) | B (Melflufen+Daratumumab+Dex) 40 mg (N=27)
Fatigue (General disorders) | 5 | 2 | 2 | 11
Asthenia (General disorders) | 4 | 1 | 2 | 7
Pyrexia (General disorders) | 2 | 1 | 1 | 6
Oedema peripheral (General disorders) | 1 | 1 | 2 | 3
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 8 | 6 | 17
Neutropenia (Blood and lymphatic system disorders) | 11 | 7 | 6 | 17
Anaemia (Blood and lymphatic system disorders) | 10 | 6 | 5 | 16
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 1 | 9
Nausea (Gastrointestinal disorders) | 4 | 2 | 0 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 5
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 4 | 6
Urinary tract infection (Infections and infestations) | 3 | 1 | 3 | 3
Infection (Infections and infestations) | 4 | 3 | 3 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 3
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 3
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3 | 1
Erythema migrans (Infections and infestations) | 0 | 0 | 2 | 0
COVID-19 (Infections and infestations) | 2 | 2 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 3 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 6
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 3
Weight decreased (Investigations) | 1 | 1 | 0 | 2
C-reactive protein increased (Investigations) | 1 | 2 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 4 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 6
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 3 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 6
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 3 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 2 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 2
Device dislocation (Product Issues) | 0 | 0 | 0 | 1
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Withdrawal syndrome (General disorders) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 1
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Bacteriuria (Infections and infestations) | 1 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 1 | 0 | 0 | 0
Carbuncle (Infections and infestations) | 1 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis clostridal (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster oticus (Infections and infestations) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Periodonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 0 | 1 | 0
Pustule (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0 | 0
Gamm-glutamyltransferase decreased (Investigations) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin fragility (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 2
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1
Cataract nuclear (Eye disorders) | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Eye oedema (Eye disorders) | 0 | 0 | 0 | 1
Scleral haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thrombosis in device (Product Issues) | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
On 04 November 2021, the study was terminated early during Phase 2a.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT03481556/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT03481556/SAP_001.pdf